CLINICAL TRIAL: NCT00001309
Title: Pharmacokinetics and Biodistribution of Ascorbic Acid in Healthy Human Subjects
Brief Title: The Body's Affect on Vitamin C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 920033; 92-DK-0033
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Biodistribution; Ascorbic Acid
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetics and Biodistribution of Ascorbic Acid (Other): Outpatient subjects will be encouraged to consume vitamin C in foods. As inpatients, vitamin C deficiency will be induced by placing subjects on a tightly restricted scorbutic diet. Plasma vitamin C will be monitored several times per week. When subjects have achieved a plasma ascorbate concentration of 5-10 micromolar, blood sampling and urine collection over 24 hours will be performed. After platelets and leukocytes are collected, ascorbate repletion will begin. Escalating doses of ascorbate will be administered orally and intravenously for the remainder of their inpatient admission. Total daily doses of 30mg, 60mg, 100mg, 200mg, 400mg, 1000mg and 2500mg will be given in two divided doses. Bioavailability of ascorbate will be determined at each dosage increment. When plasma ascorbate concentration reaches steady state for each dose, subjects will undergo 36 hr plasma sampling and a timed 48 hr urine collection.
  Interventions: Other: Vitamin C

INTERVENTIONS:
Other: Vitamin C — Outpatient subjects will be encouraged to consume vitamin C in foods. As inpatients, vitamin C deficiency will be induced by placing subjects on a tightly restricted scorbutic diet. Plasma vitamin C will be monitored several times per week. When subjects have achieved a plasma ascorbate concentration of 5-10 micromolar, blood sampling and urine collection over 24 hours will be performed. After platelets and leukocytes are collected, ascorbate repletion will begin. Escalating doses of ascorbate will be administered orally and intravenously for the remainder of their inpatient admission. Total daily doses of 30mg, 60mg, 100mg, 200mg, 400mg, 1000mg and 2500mg will be given in two divided doses. Bioavailability of ascorbate will be determined at each dosage increment. When plasma ascorbate concentration reaches steady state for each dose, subjects will undergo 36 hr plasma sampling and a timed 48 hr urine collection.

SUMMARY:
Pharmacokinetics is the term used for how the body affects a drug once it is taken. Vitamin C, also known as ascorbic acid, is an essential water soluble vitamin. Meaning, the body does not make Vitamin C it must be taken in through the diet. In this study researchers will attempt to determine how the amount of water consumed affects the level of vitamin C in the blood (specifically the plasma component of the blood).

In this study researchers will take 13 subjects and place them on a Vitamin C restricted diet. Vitamin C levels will be measured twice a week on an outpatient basis until all subjects reach a desired low level of Vitamin C (12-15 micromolar plasma ascorbic acid concentration). Subjects will then be admitted and undergo 24 hour blood and urine collection. Following the collection of samples, subjects will then begin to receive Vitamin C orally (by mouth) and intravenously (injected into the vein). The dosage of Vitamin C will gradually increase from 30 mg-2500 mg divided into two daily doses. Blood and urine samples will be collected each time the dose is increased. The study will take approximately 18 weeks after which the subjects will be discharged in healthy condition.

DETAILED DESCRIPTION:
Vitamin C (ascorbic acid, ascorbate) is an essential water soluble vitamin. Our studies at NIH were the first to demonstrate in healthy men and women how changes in a vitamin concentration in human plasma vary as a direct function of the amount ingested, over a wide range. ln the present study, we plan to achieve a prescorbutic vitamin C plasma concentration of approximately 5-10 micromolar in healthy human volunteers. We will gradually replete these subjects with incremental doses of vitamin C to measure how their plasma, red blood cell, and leukocyte concentrations will change as a function of the dose. We will also determine whether changes in vitamin C concentration result in changes in gene expression and metabolic profiles (metabolomics, lipidomics, proteomics).

Outpatient subjects will be encouraged to consume vitamin C in foods. As inpatients, vitamin C deficiency will be induced by placing subjects on a tightly restricted scorbutic diet. Plasma vitamin C will be monitored several times per week. When subjects have achieved a plasma ascorbate concentration of 5-10 micromolar, blood sampling and urine collection over 24 hours will be performed. After platelets and leukocytes are collected, ascorbate repletion will begin. Escalating doses of ascorbate will be administered orally and intravenously for the remainder of their inpatient admission. Total daily doses of 30mg, 60mg, 100mg, 200mg, 400mg, 1000mg and 2500mg will be given in two divided doses. Bioavailability of ascorbate will be determined at each dosage increment. When plasma ascorbate concentration reaches steady state for each dose, subjects will undergo 36 hr plasma sampling and a timed 48 hr urine collection. At steady state of each of 4 to 5 doses, an apheresis procedure will be performed for collection of platelets and leukocytes. lt is anticipated subjects will be discharged in healthy condition after 20-26 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 10 Males - ages 18 - 35 yrs
* 10 Females - ages 18 - 35 yrs

No more than 4 subjects during any period will remain as inpatients on the endocrine/metabolic ward. These subjects will be normal volunteers selected from colleges/universities who will:

1. Spend within a fall or spring semester (approximately 20-26 weeks) as an inpatient resident on the endocrine-metabolic ward at NIH.
2. Be willing to adhere to an ascorbate restricted diet for the duration of the time spent in the study as an inpatient at NlH.
3. Have veins adequate for venipunctures and be willing to undergo venipunctures approximately two to three times per week.
4. Refrain from ingestion of any medication and cigarette smoking and ethanol.
5. Be able to give informed consent.

EXCLUSION CRITERIA:

1. Subject non-compliance with restricted diet.
2. Pregnancy as determined by history, physical exam and urine b-HCG.
3. History of diabetes mellitus, bleeding disorders, kidney stones, glucose-6- phosphate dehydrogenase deficiency, family history of hemochromatosis/iron overload.
4. Platelet count <150,000/ul blood; prothrombin time/partial thromboplastin time (PT/PTT) > 1 second above normal upper limit.
5. Positive test for exposure to human immunodeficiency virus.
6. Positive tests for hepatitis B surface antigen, core antibody or surface antibody.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 1997-01-23 (Actual); Primary Completion 1999-08-25 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Changes in ascorbic acid concentrations | 5 years
  In this study researchers will attempt to determine how the amount of water consumed affects the level of vitamin C in the blood (specifically the plasma component of the blood).

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Levine, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1992-DK-0033.html